CLINICAL TRIAL: NCT07023861
Title: The Exploration of Novel Radionuclide-labeled HER2-targeting Antibodies in the Diagnosis of HER2-positive Malignancies
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: Affiliated Hospital of Jiangnan University (Other)
Responsible Party: Principal Investigator, Chunjing Yu, Director, Affiliated Hospital of Jiangnan University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: LS2024583
Record Dates: First submitted 2025-05-12; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer; Gastric Cancer (GC); Urothelial Carcinoma (UC)
Keywords: breast cancer; Gastric Cancer (GC); Urothelial carcinoma (UC); HER2; PET/CT; 89Zr
MeSH Terms: conditions — Breast Neoplasms; Stomach Neoplasms; Carcinoma, Transitional Cell | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 89Zr-LNCab190 (Experimental): 89Zr-LNCab190 injection (1-3 mCi) was injected intravenously for 45-60s.
  Interventions: Drug: 18F-FDG; Drug: 89Zr-LNCab190
- 89Zr-LNCab002 (Experimental): 89Zr-LNCab002 injection (1-3 mCi) was injected intravenously for 45-60s.
  Interventions: Drug: 18F-FDG; Drug: 89Zr-LNCab002
- 89Zr-LNCab072 (Experimental): 89Zr-LNCab072 injection (1-3mCi) was injected intravenously for 45-60s.
  Interventions: Drug: 18F-FDG; Drug: 89Zr-LNCab072
- 18F-FDG (Active Comparator): The corresponding patients underwent HER2 PET/CT examination within one week before and after routine 18F-FDG PET/CT imaging (control examination). PET/CT whole body scan was performed 45 min-1 h after intravenous injection of the developer, and the image processing was as usual.
  Interventions: Drug: 89Zr-LNCab190; Drug: 89Zr-LNCab002; Drug: 89Zr-LNCab072

INTERVENTIONS:
Drug: 18F-FDG — 18F-FDG is administered through a superficial dorsal vein, and the patient is given a dose of about 0.1-0.15 mCi/kg.
  Arms: 89Zr-LNCab002; 89Zr-LNCab072; 89Zr-LNCab190
Drug: 89Zr-LNCab190 — 89Zr-LNCab190 is administered through a superficial dorsal vein, and the patient is given a dose of about 1-3 mCi
  Arms: 18F-FDG; 89Zr-LNCab190
Drug: 89Zr-LNCab002 — 89Zr-LNCab002 is administered through a superficial dorsal vein, and the patient is given a dose of about 1-3 mCi
  Arms: 18F-FDG; 89Zr-LNCab002
Drug: 89Zr-LNCab072 — 89Zr-LNCab072 is administered through a superficial dorsal vein, and the patient is given a dose of about 1-3 mCi
  Arms: 18F-FDG; 89Zr-LNCab072

SUMMARY:
The purpose of this study is to develop and clinically evaluate 89Zr-labeled HER2-targeted antibodies in diagnosis and screening of HER2-positive cancer patients.

DETAILED DESCRIPTION:
Main objectives:

* Application of novel radionuclide-labeled HER2-targeting antibodies (89Zr-LNCab002, 89Zr-LNCab072, 89Zr-LNCab190) in the early diagnosis of breast cancer, gastric cancer, urothelial carcinoma and other diseases;
* To evaluate the efficacy, safety and dosimetry of 89Zr-LNCab002, 89Zr-LNCab072, 89Zr-LNCab190 in clinical PET imaging applications.

Secondary Objectives:

* To investigate the biodistribution of 89Zr-LNCab002, 89Zr-LNCab072 and 89Zr-LNCab190 in patients with breast cancer, gastric cancer and urothelial carcinoma, including the distribution of primary and metastatic tumors and normal tissues, through the evaluation of whole-body imaging and SUV values using PET/CT imaging.
* Compared with 18F-FDG, the clinical application value and diagnostic advantages of the novel radionuclide-labeled HER2-targeting antibodies 89Zr-LNCab002, 89Zr-LNCab072 and 89Zr-LNCab190 were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily signed the informed consent form and was able to complete the trial according to the protocol requirements ;
* 18-75 years old, male or female ;
* Clinical diagnosed with gastric cancer, breast cancer, urothelial carcinoma, diagnostic criteria refer to biopsy, and HER2 immunohistochemistry result is positive ;
* Presence of at least one measurable lesion in the subject's body, which can be accurately and continuously measured by the modified RECIST criteria (version 1.1) ;
* ECOG score of 0-3 ;
* Complete blood count, coagulation function and liver and kidney function meet the following criteria (no blood transfusion, no use of hematopoietic stimulating factor drugs and no use of liver protection drugs within 14 days before administration): a) Blood routine: white blood cell count (WBC) ≥ 2.5×109/L or neutrophil count (ANC) ≥1.5×109/L, platelet count (PLT) ≥ 100×109/L, hemoglobin ≥ 90 g/L; b) Coagulation function: prothrombin time (PT) or activated partial thromboplastin time (aPTT) ≤1.5×ULN (limited to patients who are not receiving anticoagulant therapy; Patients receiving anticoagulant therapy should be on a stable dose of anticoagulant); c) Liver function: total bilirubin ≤ 1.5× ULN, ALT/AST ≤ 2.5× ULN, ALP ≤ 2.5×ULN; d) Renal function: urea (UREA) ≤ 1.5×ULN, serum creatinine ≤ 1.5× ULN, creatinine clearance ≥ 50 mL/min (Cockcroft-Gault formula) ;
* Female subjects of childbearing potential must have a negative pregnancy test ;
* Female subjects of childbearing potential as well as male subjects of childbearing potential must agree to use effective contraception or restrict sexual behavior for the duration of the study ;

Exclusion Criteria:

* Those who are not suitable for PET/CT examination or cannot complete PET/CT examination for special reasons, including but not limited to claustrophobia, radiophobia, etc ;
* Those who cannot tolerate intravenous administration (such as history of needle sickness and blood sickness) ;
* Known allergy to chimeric or human antibodies or fusion proteins, or other excipients
* Presence of any of the following: a) brain metastases (except for primary or metastatic brain tumors that are asymptomatic and do not require treatment); b) carcinomatous meningitis; c) diabetes mellitus with poor glycemic control; d) Myocardial infarction within 6 months prior to screening; e) unstable angina; f) Have a previous uncontrollable cardiac arrhythmia or are currently at high risk; g) Prior coronary artery bypass grafting; h) Cerebrovascular accident within 6 months prior to screening; i) congestive heart failure (cardiac function class III-IV); j) pulmonary embolism; k) deep vein thrombosis) concomitant infection requiring intravenous antibiotic treatment within 2 weeks prior to screening; m) History of immunosuppressant therapy after organ transplantation ;
* Those who have had or are currently concomitant with primary central nervous system tumors ;
* Those with a history of acute or subacute intestinal obstruction, or inflammatory bowel disease ;
* Toxicity from prior anticancer therapy has not recovered to grade 0 or 1 (CTCAE version 5.0), with the exception of alopecia ;
* Presence of active autoimmune disease, or history of autoimmune disease requiring treatment with systemic hormones and/or immunosuppressants, or syndrome requiring systemic steroids or immunosuppressive medications;
* Received or planned to receive immune checkpoint blockade therapy, including anti-CTLA-4, anti-PD-1 or anti-PD-L1 therapeutic antibodies, within 1 year prior to screening, prior to completion of the study imaging procedure, etc ;
* Any psychiatric illness (e.g., alcohol or drug abuse, dementia, or altered mental status), or any other condition that affects study compliance, impairs the patient's ability to understand informed consent, or in the opinion of the investigator, would cause the patient to be unable to participate in the study or interfere with the interpretation of the study results ;
* Those who have participated in clinical trials of radiopharmaceuticals within 1 month prior to screening ;
* Drugs/clinical operators who have been evaluated by the investigator within 1 month prior to screening to affect the uptake of 89Zr-LNCab002, 89Zr-LNCab190 and 89Zr-LNCab072;
* Patients who did not meet the requirements as assessed by the investigator.

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-07 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Tumor Uptake Value (SUVmax) of HER2-Targeted PET/CT Compared with 18F-FDG PET/CT | Day 1 post-injection
  The maximum standardized uptake value (SUVmax) of identified lesions on HER2-targeted PET/CT using 89Zr-LNCab190, 89Zr-LNCab002, and 89Zr-LNCab072 will be measured and compared with the SUVmax of lesions detected on 18F-FDG PET/CT imaging in the same patients.
  Units of Measure: SUVmax (unitless)
Number of Lesions Detected by HER2-Targeted PET/CT Compared with 18F-FDG PET/CT | Day 1 post-injection
  The number of lesions detected by HER2-targeted PET/CT using 89Zr-labeled antibodies will be recorded and compared to the number of lesions detected by 18F-FDG PET/CT imaging in the same patient population.
  Units of Measure: Number of lesions

SECONDARY OUTCOMES:
Biodistribution of 89Zr-Labeled HER2-Targeted Antibodies in Normal Organs | Day 1 post-injection
  The biodistribution of 89Zr-LNCab190, 89Zr-LNCab002, and 89Zr-LNCab072 will be evaluated by measuring the mean standardized uptake values (SUVmean) in various normal organs (e.g., liver, kidney, lung, spleen, bone marrow) during HER2-targeted PET/CT imaging.
  Units of Measure: SUVmean (unitless)

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu, China